CLINICAL TRIAL: NCT04293796
Title: Refusal of Breast Surgery in Patients With Breast Cancer With a Clinical Complete Response (cCR) After Neoadjuvant Systemic Therapy and a Confirmed Pathological Complete Response (pCR) Using Vacuum-assisted Biopsy (VAB) and Sentinel Lymph Node Biopsy (SLNB)
Acronym: VAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PetrovRIO
Record Dates: First submitted 2020-01-19; First posted 2020-03-03 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Refusal of Breast Surgery in Patients With Breast Cancer With a cCR After NST and a Confirmed Pathological Complete Response (pCR) Using VAB and SLNB
MeSH Terms: conditions — Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TNBC group (Experimental): A group with TNBC in neoadjuvant therapy will receive 4 cycles of neoadjuvant polychemotherapy according to the AC regimen (doxorubicin 60 mg / m2, cyclophosphamide 600 mg / m2) once every 21 days, then 12 cycles of neoadjuvant polychemotherapy according to the paclitaxel 60-100 mg / m² scheme in 1 day + carboplatin AUC 2 1 p in 7 days. VAB with SLNB and radiation therapy on the remaining breast tissue with cCR and pCR patients. Patients with residual breast cancer undergo standart surgery procedure.
  Interventions: Procedure: Vacuum-assisted biopsy
- HER2-positive breast cancer group (Experimental): ER + - / HER2 + will receive 4 cycles of neoadjuvant polychemotherapy according to the AC regimen (doxorubicin 60 mg / m2, cyclophosphamide 600 mg / m2) once every 21 days, then docetaxel 75-100 mg / m² on the 1st day + trastuzumab 6 mg / kg (loading dose of 8 mg / kg) on the 1st day + pertuzumab 420 mg (loading dose of 840 mg) on the 1st day; 4 cycles, 1 time in 21 days and surgical treatment. In adjuvant therapy, a group of patients with HER2-positive breast cancer will receive trastuzumab for up to one year and hormone therapy with an antiestrogen (tamoxifen) or aromatase inhibitors in ER + / HER2 + tumors. VAB with SLNB and radiation therapy on the remaining breast tissue with cCR and pCR patients. Patients with residual breast cancer undergo standart surgery procedure.
  Interventions: Procedure: Vacuum-assisted biopsy

INTERVENTIONS:
Procedure: Vacuum-assisted biopsy — The vacuum-assisted (7-10G), minimal invasive biopsy (VAB), either guided by ultrasound, after neoadjuvant systemic treatment on patients with clinical complete response on primary breast cancer management we recommend to take at least 12 biopsies with 7-10G needle sizes with sentinel lymph node biopsy.

SUMMARY:
The main goal of the study is to abandon breast surgery in patients with breast cancer with a clinical complete response (cCR) after neoadjuvant systemic therapy and confirmed pCR using Vacuum-assisted biopsy (VAB) and sentinel lymph node biopsy (SLNB).

Evidence of the high diagnostic accuracy (sensitivity and specificity) of vacuum aspiration biopsy in determining pCR in patients with clinical complete response after neoadjuvant systemic therapy will allow abandoning breast surgery in favor of radiation therapy alone, improving the quality of life of these patients.

DETAILED DESCRIPTION:
Vacuum-assisted removal and biopsy of the tumor bed after neoadjuvant systemic therapy (NST) in patients with clinical complete clinical response with a biopsy of sientinel lymph nodes is in the future a modern alternative to the standard, often crippling and traumatic surgical procedures and does not require additional financial costs for the reconstruction of the breast.

There are only two trial visits that are specific to the trial. All other visits will be routine visits.

The first trial visit before NST will take place in order to provide the patient with detailed information on the study, its' aims, the VAB procedure, and its risks. The patient will be asked to sign a form of informed consent.

In the second visit after the NST, VAB planning will be carried out. This visit may vary depending on the patient, the tumor, and the characteristics of the study site. We will provide each test participant with the opportunity to choose the appropriate conditions for the procedure.

The VAB procedure with a sentinel lymph node biopsy will be performed in the operating room Research objectives

1. To evaluate the frequency of coincidence of the clinical complete or partial response (cCR and PR) with pathological complete response (pCR).
2. To study the frequency of detecting a residual tumor in the mammary gland using a Vacuum-assisted biopsy or another type of core biopsy and / or detection of metastases in regional lymph nodes (sentinel lymph node biopsy) in comparison with a standard pathological study of the surgical material and regional (including sentinel ) lymph nodes.
3. To analyze the frequency of false-positive conclusions of a vacuum aspiration biopsy of the tumor bed about the achievement of pathological complete response (pCR) in comparison with a standard pathological study of a surgical material.
4. To study the long-term results (local-regional relapse, survival) of surgical treatment of patients with clinical complete response (cCR) after neoadjuvant systemic therapy, including residual disease compared with patients who achieved pathological complete response (pCR).
5. To develop an algorithm for treating patients with clinical complete response, with a confirmed pathological complete response using a tumor bed biopsy and targeted biopsy of sentinel lymph nodes (taking into account the initial characteristics: age, stage with TNM, disease subtypes, the presence of a genetic mutation BRCA1 / 2).

Ultrasound guided VAB will be performed on breast cancer patients with clinical complete response (cCR) after NST.

The pathological results of the VAB specimen will be generally categorized as follows:

1. Residual tumor cells in VAB specimen (=non-pCR)
2. No residual tumor cells in the VAB specimen and VAB representative of former tumor region (="pCR in VAB")
3. No residual tumor cells in the VAB specimen but VAB unclear or not representative of former tumor region (=possible sampling error). These VABs are categorized as uninformative for the primary endpoint of the clinical trial.

The results will be compared with the results of a pathological examination of a surgical material.

ELIGIBILITY:
Inclusion Criteria:

Triple negative breast cancer / HER2-positive breast cancer (ER / PR +/-)

* age> 18 years.
* morphologically confirmed diagnosis of breast cancer, IIA-IIIA stage
* ECOG score 0-1.
* life expectancy of more than 3 months.
* the consent of patients to use reliable methods of contraception throughout the study
* adequate liver and bone marrow function
* the absence of contraindications to surgical intervention (including anesthetic risk is taken into account).

Exclusion Criteria:

* Inconsistency with inclusion criteria.
* Conducting earlier any systemic therapy for breast cancer.
* stage 4 cancer
* carrier mutations of the BRCA1 / 2 gene
* severe uncontrolled concomitant chronic diseases or acute diseases
* the presence of a second malignant tumor
* pregnancy or lactation
* acute conditions and complications, which, according to the doctor, interfere with treatment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
False negative rate of vacuum-assisted biopsy (FNR) | During the surgery
  Achieving a false-negative rate (FNR) of less than 15% in the surgical and vacuum-assisted biopsy specimens

CONTACTS AND LOCATIONS:
Overall Officials: Petr Krivorotko, MD,PhD, Principal Investigator — N.N. Petrov Research Institute of Oncology; Vladimir Semiglazov, Professor, Study Director — N.N.Petrov Research Institute of Oncology
Locations (1):
- Petr Krivorotko, Saint Petersburg, Russia